CLINICAL TRIAL: NCT03229967
Title: Gastrointestinal Microbiota Influence on the Pathogenesis of Bronchopulmonary Dysplasia in Very Low Birthweight Neonates
Brief Title: Gastrointestinal Microbiome Influence on the Development of Bronchopulmonary Dysplasia
Acronym: MiBPD
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Principal Investigator, Kent Avery Willis, MD, Neonatal-Perinatal Medicine Fellow, University of Tennessee
Other Study IDs: 17-05311-XP
Record Dates: First submitted 2017-07-11; First posted 2017-07-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary dysplasia; Microbiome; Microbiota; Premature infant; Observational cohort study
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal Stool Sample (contains bacterial and fungal DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exploration Cohort: Up to 150 VLBW (very low birthweight) infants enrolled from the Regional One Health NICU (neonatal intensive care unit). Weekly stool samples will be obtained. After 36 weeks infants diagnosed with BPD per NIH guidelines, will be matched with infants without BPD. Stool samples from these infants will be sent for 16s rRNA (ribosomal ribonucleic acid) sequencing after conclusion of initial enrollment period. ITS (internal transcribed spacer) DNA may also be used to characterize fungal communities.
  Interventions: Diagnostic Test: 16S rRNA stool microbiome sequencing.
- Validation Cohort: Up to 10 VLBW infants enrolled from the Le Bonheur Children's Hospital NICU. Weekly stool samples will be obtained. After 36 weeks infants diagnosed with BPD per NIH guidelines willl be matched with infants without BPD. Stool samples from these infants will be sent for 16s rRNA sequencing after conclusion of initial enrollment period.
  Interventions: Diagnostic Test: 16S rRNA stool microbiome sequencing.
- Well Baby Cohort: 40 Well Baby Infants have been enrolled and may be used for secondary analysis of microbial community composition of the meconium.
  Interventions: Diagnostic Test: 16S rRNA stool microbiome sequencing.

INTERVENTIONS:
Diagnostic Test: 16S rRNA stool microbiome sequencing. — This is an observational cohort that will undergo gut microbiome sequencing.

SUMMARY:
The purpose of this study is to advance our knowledge of the factors that contribute to the development of bronchopulmonary dysplasia (BPD), a chronic lung affecting premature infants. Specifically, the investigators will determine the complexity of the gut microbiota, the genera of the bacteria that naturally live in the gut, and determine if the relative diversity of the gut bacteria is a prognostic indicator of BPD. To accomplish this, the investigators propose to characterize the microbiota of human premature newborns with BPD, then validate this potential mechanism in mice. The investigators will enroll very low birthweight premature infants admitted to the neonatal intensive care units (NICU) at Le Bonheur Children's Hospital and Regional One Health that are at high risk to develop BPD. A cohort of well full term newborns will also be enrolled. Non-invasive stool samples will be obtained weekly over the first month of life. Infants that eventually develop BPD will be paired with infants that did not develop BPD. Stool samples from these infants will be sent for analysis. The investigators expect that reduced complexity of the gut microbiome is associated with BPD. The investigators will model the contribution of reduced microbiome complexity to the risk to develop BPD or death, as well as the association with disease severity. The project investigates important factors leading to the development of BPD, and has the potential to directly translate to therapy for the most significant pulmonary complication of prematurity.

ELIGIBILITY:
Inclusion Criteria:

1. Newborn humans less than 1 week of age with a birthweight less than 1,500 g, or fetuses with impending delivery and estimated birthweight of less than 1,500 grams. No individuals will be excluded on the basis of sex or ethnicity.
2. Parents can understand and comply with planned study procedures.
3. Parents provide assent/permission prior to any study procedures.

Inclusion criteria mothers:

1. The mother's of infants meeting the infant inclusion criteria above.

Exclusion Criteria:

1. Diagnosed immunodeficiency disorder.
2. Currently receiving investigational immunomodulatory, probiotic or antiviral agent.
3. Infants whose mothers meet the exclusion criteria below.

Exclusion criteria mothers:

1. Diagnosed immunodeficiency disorder
2. Currently receiving investigational immunomodulatory, probiotic or antiviral agents
3. Lacking the mental capacity (e.g. due to pain, anesthesia, mental impairment) to provide informed consent for themselves or assent for the participation of their infant.
4. Having an infant that meets the infant exclusion criteria.

Ages: 0 Days to 7 Days | Sex: All
Age Groups: Child
Study Population: Study Population will be composed of VLBW infants (birthweight less than 1500 grams) and their mothers (Including 40 term infants and their mothers)
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia (BPD) | 36 weeks corrected gestational age, until the date of death or initial hospital discharge whichever occurs first, assessed up to up to 3 months
  National Institute of Child Health and Disease (NICHD) consensus definition
Death | from the date of enrollment until the date of death or initial hospital discharge, whichever occurs first, assessed up to up to 3 months

SECONDARY OUTCOMES:
Necrotizing Enterocolitis (NEC) | from the date of enrollment until the date of initial hospital discharge or death, whichever occurs first, assessed up to up to 3 months
  Modified Bell's staging for NEC > Stage 2
Maternal Chorioamnionitis | presence on admission

OTHER OUTCOMES:
Maternal perinatal antibiotic exposure | from hospital admission until birth of infant
Infant antibiotic exposure | birth until 36 weeks corrected gestational age

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Regional One Health, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
MiSeq data will be placed in a public repository

REFERENCES:
- [Result] Willis KA, Purvis JH, Myers ED, Aziz MM, Karabayir I, Gomes CK, Peters BM, Akbilgic O, Talati AJ, Pierre JF. Fungi form interkingdom microbial communities in the primordial human gut that develop with gestational age. FASEB J. 2019 Nov;33(11):12825-12837. doi: 10.1096/fj.201901436RR. Epub 2019 Aug 31. PMID 31480903

DOCUMENTS (1):
  • Informed Consent Form (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03229967/ICF_000.pdf